CLINICAL TRIAL: NCT02545049
Title: A Randomized, Double-blind, Placebo-controlled, Parallel-group, Multicenter, Event-driven Phase 3 Study to Investigate Efficacy and Safety of Finerenone on the Reduction of Cardiovascular Morbidity and Mortality in Subjects With Type 2 Diabetes Mellitus and the Clinical Diagnosis of Diabetic Kidney Disease in Addition to Standard of Care.
Brief Title: Efficacy and Safety of Finerenone in Subjects With Type 2 Diabetes Mellitus and the Clinical Diagnosis of Diabetic Kidney Disease
Acronym: FIGARO-DKD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 17530; 2015-000950-39 (EudraCT Number)
Record Dates: First submitted 2015-09-02; First posted 2015-09-09 (Estimated); Results first posted 2022-04-15 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: Diabetic Kidney Disease
Keywords: Type 2 Diabetes; Kidney diseases
MeSH Terms: conditions — Diabetic Nephropathies; Diabetes Mellitus, Type 2; Kidney Diseases | interventions — finerenone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BAY94-8862 (Experimental): Finerenone tablet
  Interventions: Drug: Finerenone (BAY94-8862)
- Placebo (Placebo Comparator): Matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Finerenone (BAY94-8862) — 10 mg or 20 mg Finerenone tablet to be given orally, once daily.
  Arms: BAY94-8862
Drug: Placebo — Matching placebo to be taken orally, once daily.
  Arms: Placebo

SUMMARY:
The purpose of this study was to evaluate whether oral finerenone (study drug), in addition to standard daily therapy, is effective and safe in treating patients with type 2 diabetes mellitus and diabetic kidney disease, when compared to a placebo.

ELIGIBILITY:
Inclusion Criteria:

* Men or women ≥18 years of age
* Subjects with Type Type 2 Diabetes Mellitus as defined by the American Diabetes Association
* Diagnosis of Diabetic Kidney Disease with persistent high albuminuria or persistent very high albuminuria at the Run-In and Screening Visit
* Pretreated with either angiotensin-converting enzyme inhibitor (ACEI) or angiotensin receptor blocker (ARB) at maximal tolerated labeled dose without adjustments
* Serum potassium <=4.8 mmol/L

Exclusion Criteria:

* Confirmed significant non-diabetic renal disease, including clinically relevant renal artery stenosis
* Uncontrolled arterial hypertension (ie, mean sitting systolic blood pressure (SBP) ≥170 mmHg or mean sitting diastolic blood pressure(DBP) ≥110 mmHg at run in visit, or mean sitting SBP ≥160 mmHg or mean sitting DBP ≥100 mmHg at screening)
* Clinical diagnosis of chronic heart failure with reduced ejection fraction (HFrEF) and persistent symptoms {New York Heart Association (NYHA) class II - IV} at Run in visit [class 1A recommendation for mineralcorticoid receptor antagonist (MRAs)]
* Dialysis for acute renal failure within 12 weeks of Run-in visit
* Renal allograft in place or scheduled kidney transplant within next 12 months
* Glycated hemoglobin (HbA1c) >12%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7352 (Actual)
Dates: Start 2015-09-17 (Actual); Primary Completion 2021-02-02 (Actual); Study Completion 2021-02-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (701):
- United States (127):
  - Birmingham, Alabama
  - Fort Payne, Alabama
  - Huntsville, Alabama
  - Mesa, Arizona
  - Phoenix, Arizona
  - Prescott, Arizona
  - Tucson, Arizona
  - Bakersfield, California
  - Chula Vista, California
  - Dublin, California
  - El Centro, California
  - Fresno, California
  - La Mesa, California
  - Loma Linda, California
  - Los Angeles, California
  - Northridge, California
  - Port Hueneme, California
  - Poway, California
  - Rancho Cucamonga, California
  - Rialto, California
  - Roseville, California
  - San Diego, California
  - Santa Rosa, California
  - Torrance, California
  - Vista, California
  - New Haven, Connecticut
  - Waterbury, Connecticut
  - Fort Lauderdale, Florida
  - Hialeah, Florida
  - Hollywood, Florida
  - Jacksonville, Florida
  - Miami, Florida
  - Miami Beach, Florida
  - Miami Gardens, Florida
  - Miami Lakes, Florida
  - New Port Richey, Florida
  - Ocala, Florida
  - Orlando, Florida
  - Palm Harbor, Florida
  - Sarasota, Florida
  - Tampa, Florida
  - West Palm Beach, Florida
  - Winter Haven, Florida
  - Atlanta, Georgia
  - Augusta, Georgia
  - Lawrenceville, Georgia
  - Macon, Georgia
  - Honolulu, Hawaii
  - Chicago, Illinois
  - Elgin, Illinois
  - Morton, Illinois
  - Springfield, Illinois
  - Indianapolis, Indiana
  - Iowa City, Iowa
  - West Des Moines, Iowa
  - Hutchinson, Kansas
  - Topeka, Kansas
  - Wichita, Kansas
  - Metairie, Louisiana
  - Monroe, Louisiana
  - New Orleans, Louisiana
  - Shreveport, Louisiana
  - Boston, Massachusetts
  - Ann Arbor, Michigan
  - Flint, Michigan
  - Kalamazoo, Michigan
  - Minneapolis, Minnesota
  - Columbia, Missouri
  - Jefferson City, Missouri
  - Kansas City, Missouri
  - St Louis, Missouri
  - Omaha, Nebraska
  - Las Vegas, Nevada
  - Reno, Nevada
  - Newark, New Jersey
  - Albuquerque, New Mexico
  - Albany, New York
  - Brooklyn, New York
  - New York, New York
  - Rosedale, New York
  - Smithtown, New York
  - Staten Island, New York
  - Asheboro, North Carolina
  - Chapel Hill, North Carolina
  - Charlotte, North Carolina
  - Greenville, North Carolina
  - New Bern, North Carolina
  - Winston-Salem, North Carolina
  - Canton, Ohio
  - Willoughby Hills, Ohio
  - Beaver, Pennsylvania
  - Bethlehem, Pennsylvania
  - Hershey, Pennsylvania
  - Jersey Shore, Pennsylvania
  - Anderson, South Carolina
  - Charleston, South Carolina
  - Greenville, South Carolina
  - Murrells Inlet, South Carolina
  - Myrtle Beach, South Carolina
  - Orangeburg, South Carolina
  - Chattanooga, Tennessee
  - Memphis, Tennessee
  - Nashville, Tennessee
  - Arlington, Texas
  - Corpus Christi, Texas
  - Dallas, Texas
  - El Paso, Texas
  - Houston, Texas
  - Kingwood, Texas
  - McAllen, Texas
  - McKinney, Texas
  - Missouri City, Texas
  - Pearland, Texas
  - Pflugerville, Texas
  - San Antonio, Texas
  - Sugar Land, Texas
  - Tomball, Texas
  - Waco, Texas
  - Salt Lake City, Utah
  - Burlington, Vermont
  - Alexandria, Virginia
  - Charlottesville, Virginia
  - Manassas, Virginia
  - Salem, Virginia
  - Virginia Beach, Virginia
  - Spokane, Washington
  - Tacoma, Washington
- Argentina (10):
  - CABA, Buenos Aires
  - Junín, Buenos Aires
  - Lanús, Buenos Aires
  - Mar del Plata, Buenos Aires
  - Sarandí, Buenos Aires
  - Buenos Aires, Ciudad Auton. de Buenos Aires
  - CABA, Ciudad Auton. de Buenos Aires
  - Ciudad Autón. de Buenos Aires, Ciudad Auton. de Buenos Aires
  - Córdoba
  - San Luis
- Australia (16):
  - Garran, Australian Capital Territory
  - Gosford, New South Wales
  - Kanwal, New South Wales
  - Liverpool, New South Wales
  - New Lambton Heights, New South Wales
  - Wollongong, New South Wales
  - Brisbane, Queensland
  - Adelaide, South Australia
  - Fitzroy, Victoria
  - Heidelberg, Victoria
  - Melbourne, Victoria
  - Prahran, Victoria
  - Reservoir, Victoria
  - Richmond, Victoria
  - St Albans, Victoria
  - Elizabeth Vale
- Austria (9):
  - Graz, Styria
  - Saint Stefan, Styria
  - Zams, Tyrol
  - Linz, Upper Austria
  - Feldkirch, Vorarlberg
  - Innsbruck
  - Salzburg
  - Vienna
  - Wels
- Belgium (8):
  - Bruxelles - Brussel
  - Edegem
  - Ghent
  - Ieper
  - Kortrijk
  - Leuven
  - Liège
  - Roeselare
- Brazil (15):
  - Fortaleza, Ceará
  - Brasília, Federal District
  - Aparecida de Goiânia, Goiás
  - Goiânia, Goiás
  - Juiz de Fora, Minas Gerais
  - Uberlândia, Minas Gerais
  - Campina Grande do Sul, Paraná
  - Curitiba, Paraná
  - Porto Alegre, Rio Grande do Sul
  - São Bernardo do Campo, São Paulo
  - São José do Rio Preto, São Paulo
  - São José dos Campos, São Paulo
  - São Paulo, São Paulo
  - Rio de Janeiro
  - São Paulo
- Bulgaria (14):
  - Blagoevgrad
  - Botevgrad
  - Dimitrovgrad
  - Gorna Oryahovitsa
  - Kazanlak
  - Kozloduy
  - Lukovit
  - Plovdiv
  - Razgrad
  - Sliven
  - Sofia
  - Stara Zagora
  - Varna
  - Yambol
- Canada (24):
  - Edmonton, Alberta
  - Burnaby, British Columbia
  - Coquitlam, British Columbia
  - New Westminster, British Columbia
  - Mount Pearl, Newfoundland and Labrador
  - St. John's, Newfoundland and Labrador
  - Halifax, Nova Scotia
  - Cambridge, Ontario
  - Greater Sudbury, Ontario
  - Hamilton, Ontario
  - Kitchener, Ontario
  - Newmarket, Ontario
  - Oshawa, Ontario
  - Ottawa, Ontario
  - Sarnia, Ontario
  - Smith Falls, Ontario
  - Thornhill, Ontario
  - Toronto, Ontario
  - Waterloo, Ontario
  - Greenfield Park, Quebec
  - Laval, Quebec
  - Mirabel, Quebec
  - Montreal, Quebec
  - Québec
- Chile (6):
  - Osorno, Los Lagos Region
  - Las Condes, Santiago Metropolitan
  - Providencia, Santiago Metropolitan
  - San Bernardo, Santiago Metropolitan
  - San Miguel, Santiago Metropolitan
  - Santiago
- China (32):
  - Xiamen, Fujian
  - Lanzhou, Gansu
  - Guangzhou, Guangdong
  - Zhuhai, Guangdong
  - Nanning, Guangxi
  - Haikou, Hainan
  - Wuhan, Hubei
  - Changsha, Hunan
  - Hohhot, Inner Mongolia
  - Changzhou, Jiangsu
  - Huai'an, Jiangsu
  - Lianyungang, Jiangsu
  - Nanjing, Jiangsu
  - Suzhou, Jiangsu
  - Wuxi, Jiangsu
  - Yancheng, Jiangsu
  - Nanchang, Jiangxi
  - Changchun, Jilin
  - Shenyang, Liaoning
  - Yinchuan, Ningxia
  - Xi'an, Shaanxi
  - Qingdao, Shandong
  - Taiyuan, Shanxi
  - Chengdu, Sichuan
  - Ürümqi, Xinjiang
  - Hangzhou, Zhejiang
  - Taizhou, Zhejiang
  - Wenzhou, Zhejiang
  - Beijing
  - Chongqing
  - Shanghai
  - Tianjin
- Colombia (14):
  - Medellín, Antioquia
  - Barranquilla, Atlántico
  - Bogotá, Bogota D.C.
  - Cundinamarca, Bogota D.C.
  - Manizales, Caldas Department
  - Zipaquirá, Cundinamarca
  - Pasto, Departamento de Nariño
  - Armenia, Quindío Department
  - Pereira, Risaralda Department
  - Cali, Valle del Cauca Department
  - Barranquilla
  - Bogotá
  - Floridablanca
  - Medellín
- Czechia (17):
  - Beroun
  - Brandýs nad Labem
  - Břeclav
  - Česká Lípa
  - Český Krumlov
  - Frýdek-Místek
  - Hodonín
  - Holešov
  - Hranice
  - Kopřivnice
  - Krnov
  - Mladá Boleslav
  - Olomouc
  - Ostrava
  - Pilsen
  - Prague
  - Vlašim
- Denmark (15):
  - Aalborg
  - Aarhus N
  - Esbjerg
  - Gentofte Municipality
  - Hellerup
  - Herlev
  - Hillerød
  - Holbæk
  - Holstebro
  - Hvidovre
  - Kolding
  - København NV
  - Odense C
  - Svendborg
  - Viborg
- Finland (12):
  - Jyväskylä
  - Kajaani
  - Kerava
  - Klaukkala
  - Kuopio
  - Nurmijärvi
  - Oulu
  - Rauma
  - Seinäjoki
  - Tampere
  - Turku
  - Vantaa
- France (16):
  - Bois-Guillaume
  - Boulogne-sur-Mer
  - Brest
  - Colmar
  - Dijon
  - Grenoble
  - Le Coudray
  - Le Creusot
  - Lyon
  - Mulhouse
  - Nîmes
  - Paris
  - Saint-Herblain
  - Tourcoing
  - Vandœuvre-lès-Nancy
  - Vénissieux
- Germany (27):
  - Heidelberg, Baden-Wurttemberg
  - Ludwigsburg, Baden-Wurttemberg
  - Sinzheim, Baden-Wurttemberg
  - Nuremberg, Bavaria
  - Schweinfurt, Bavaria
  - Würzburg, Bavaria
  - Elsterwerda, Brandenburg
  - Bad Homburg, Hesse
  - Bad König, Hesse
  - Frankfurt am Main, Hesse
  - Göttingen, Lower Saxony
  - Hanover, Lower Saxony
  - Bad Oeynhausen, North Rhine-Westphalia
  - Dortmund, North Rhine-Westphalia
  - Düsseldorf, North Rhine-Westphalia
  - Essen, North Rhine-Westphalia
  - Münster, North Rhine-Westphalia
  - Nettetal, North Rhine-Westphalia
  - Witten, North Rhine-Westphalia
  - Ludwigshafen am Rhein, Rhineland-Palatinate
  - Mainz, Rhineland-Palatinate
  - Dresden, Saxony
  - Leipzig, Saxony
  - Magdeburg, Saxony-Anhalt
  - Jena, Thuringia
  - Berlin
  - Hamburg
- Greece (6):
  - Alexandroupoli
  - Athens
  - Chaïdári
  - Larissa
  - Nea Ionia
  - Thessaloniki
- Hong Kong (4):
  - Hong Kong
  - Shatin
  - Sheung Wan
  - Wong Tai Sin
- Hungary (13):
  - Baja
  - Balatonfüred
  - Budapest
  - Debrecen
  - Eger
  - Kistarcsa
  - Nyíregyháza
  - Pápa
  - Siófok
  - Szeged
  - Szentes
  - Székesfehérvár
  - Szombathely
- Ireland (3):
  - Cork
  - Dublin
  - Galway
- Israel (16):
  - Afula
  - Ashkelon
  - Beersheba
  - Haifa
  - Holon
  - Jerusalem
  - Kfar Saba
  - Nahariya
  - Nazareth
  - Ramat Gan
  - Rehovot
  - Safed
  - Sakhnin
  - Tel Aviv
  - Tiberias
  - Ẕerifin
- Italy (15):
  - Napoli, Campania
  - Bologna, Emilia-Romagna
  - Parma, Emilia-Romagna
  - Reggio Emilia, Emilia-Romagna
  - Genoa, Liguria
  - Bergamo, Lombardy
  - Milan, Lombardy
  - Monza Brianza, Lombardy
  - Turin, Piedmont
  - Cagliari, Sardinia
  - Sassari, Sardinia
  - Catania, Sicily
  - Messina, Sicily
  - Pisa, Tuscany
  - Verona, Veneto
- Japan (51):
  - Nagoya, Aichi-ken
  - Toyota, Aichi-ken
  - Funabashi, Chiba
  - Ichikawa, Chiba
  - Matsuyama, Ehime
  - Chikushino-shi, Fukuoka
  - Kasuga, Fukuoka
  - Kitakyushu, Fukuoka
  - Shirakawa, Fukushima
  - Ōgaki, Gifu
  - Maebashi, Gunma
  - Higashihiroshima, Hiroshima
  - Asahikawa, Hokkaido
  - Hakodate, Hokkaido
  - Obihiro, Hokkaido
  - Sapporo, Hokkaido
  - Kobe, Hyōgo
  - Naka, Ibaraki
  - Ushiku, Ibaraki
  - Komatsu, Ishikawa-ken
  - Sanuki, Kagawa-ken
  - Takamatsu, Kagawa-ken
  - Atsugi, Kanagawa
  - Fujisawa, Kanagawa
  - Kamakura, Kanagawa
  - Yokohama, Kanagawa
  - Tamana, Kumamoto
  - Yatsushiro, Kumamoto
  - Sasebo, Nagasaki
  - Beppu, Oita Prefecture
  - Yufu, Oita Prefecture
  - Nakagami-gun, Okinawa
  - Shimajiri, Okinawa
  - Matsubara, Osaka
  - Suita, Osaka
  - Kawaguchi, Saitama
  - Sayama, Saitama
  - Ōtsu, Shiga
  - Iwata, Shizuoka
  - Oyama, Tochigi
  - Minato, Tokyo
  - Musashino, Tokyo
  - Shibuya-ku, Tokyo
  - Tacchikawa, Tokyo
  - Fukui
  - Fukuoka
  - Kagoshima
  - Kumamoto
  - Nagasaki
  - Osaka
  - Saitama
- Lithuania (4):
  - Kaunas
  - Klaipėda
  - Utena
  - Vilnius
- Malaysia (8):
  - Johor Bahru
  - Kelantan
  - Kuala Lumpur
  - Kuala Pahang
  - Kuala Selangor
  - Perak
  - Pulau Pinang
  - Putrajaya
- Mexico (15):
  - Guadalajara, Jalisco
  - Mexico City, Mexico City
  - México D.F., Mexico City
  - México, D. F., Mexico City
  - Cuernavaca, Morelos
  - Monterrey, Nuevo León
  - Querétaro City, Querétaro
  - San Juan del Río, Querétaro
  - Culiacán, Sinaloa
  - Mazatlán, Sinaloa
  - Puerto de Veracruz, Veracruz
  - Xalapa, Veracruz
  - Aguascalientes
  - Chihuahua City
  - Durango
- Netherlands (12):
  - Alkmaar
  - Almere Stad
  - Amersfoort
  - Amsterdam
  - Apeldoorn
  - Breda
  - Eindhoven
  - Geleen
  - Groningen
  - Hoogeveen
  - The Hague
  - Zwijndrecht
- New Zealand (7):
  - Auckland
  - Christchurch
  - Hamilton
  - Hawkes Bay
  - Palmerston North
  - Tauranga
  - Wellington
- Norway (9):
  - Ålesund
  - Hamar
  - Kløfta
  - Kongsvinger
  - Kristiansand
  - Levanger
  - Lierskogen
  - Oslo
  - Skedsmokorset
- Philippines (4):
  - Iloilo City
  - Marikina City
  - Pasig
  - Quezon City
- Poland (17):
  - Bialystok
  - Bydgoszcz
  - Chojnice
  - Gdansk
  - Gdynia
  - Katowice
  - Krakow
  - Lodz
  - Lublin
  - Poznan
  - Rzeszów
  - Skorzewo
  - Szczecin
  - Torun
  - Warsaw
  - Wroclaw
  - Zabrze
- Portugal (14):
  - Covilha, Castelo Branco District
  - Loures, Lisbon District
  - Funchal, Madeira
  - Matosinhos Municipality, Porto District
  - Torres Novas, Santarém District
  - Setúbal, Setúbal District
  - Almada
  - Amadora
  - Braga
  - Faro
  - Leiria
  - Lisbon
  - Porto
  - Viana do Castelo
- Puerto Rico (2):
  - Cidra
  - San Juan
- Romania (13):
  - Alba Iulia, Alba
  - Oradea, Bihor County
  - Baia Mare, Maramureş
  - Ploieşti, Prahova
  - Timișoara, Timiș County
  - Brasov
  - Bucharest
  - Cluj-Napoca
  - Galati
  - Iași
  - Oradea
  - Satu Mare
  - Timișoara
- Russia (24):
  - Arkhangelsk
  - Barnaul
  - Chelyabinsk
  - Irkutsk
  - Izhevsk
  - Kazan'
  - Kemerovo
  - Kirov
  - Krasnodar
  - Krasnoyarsk
  - Kursk
  - Moscow
  - Nizhny Novgorod
  - Novosibirsk
  - Omsk
  - Orenburg
  - Perm
  - Saint Petersburg
  - Saratov
  - Stavropol
  - Syktyvkar
  - Voronezh
  - Yaroslavl
  - Yekaterinburg
- Singapore, Singapore
- Slovakia (6):
  - Banská Bystrica
  - Bardejov
  - Nitra
  - Rimavská Sobota
  - Rožňava
  - Žilina
- South Africa (15):
  - Port Elizabeth, Eastern Cape
  - Benoni, Gauteng
  - Johannesburg, Gauteng
  - Lenasia South, Gauteng
  - Newtown, Gauteng
  - Pretoria, Gauteng
  - Soweto, Gauteng
  - Durban, KwaZulu-Natal
  - Isipingo Rail, KwaZulu-Natal
  - Tongaat, KwaZulu-Natal
  - Middelburg, Mpumalanga
  - Witbank, Mpumalanga
  - Cape Town, Western Cape
  - Somerset West, Western Cape
  - Worcester, Western Cape
- South Korea (7):
  - Wŏnju, Gang''weondo
  - Anyang-si, Gyeonggido
  - Seongnam-si, Gyeonggido
  - Seoul, Seoul Teugbyeolsi
  - Busan
  - Daegu
  - Seoul
- Spain (18):
  - Ferrol, A Coruña
  - Badalona, Barcelona
  - L'Hospitalet de Llobregat, Barcelona
  - Manresa, Barcelona
  - Sant Joan Despí, Barcelona
  - Jerez de la Frontera, Cádiz
  - Burela de Cabo, Lugo
  - Alcalá de Henares, Madrid
  - Getafe, Madrid
  - Sagunto, Valencia
  - A Coruña
  - Barcelona
  - Córdoba
  - Granada
  - Jaén
  - Madrid
  - Málaga
  - Valencia
- Sweden (7):
  - Gothenburg
  - Lund
  - Örebro
  - Rättvik
  - Skövde
  - Stockholm
  - Uppsala
- Switzerland (5):
  - Olten, Canton of Solothurn
  - Sankt Gallen, Canton of St. Gallen
  - Lausanne, Canton of Vaud
  - Bern
  - Geneva
- Taiwan (6):
  - Changhua
  - Kaohsiung City
  - New Taipei City
  - Taichung
  - Taipei
  - Taoyuan District
- Thailand (3):
  - Bangkok
  - Chiang Mai
  - Khon Kaen
- Turkey (Türkiye) (9):
  - Ankara
  - Antalya
  - Aydin
  - Istanbul
  - Izmir
  - Kayseri
  - Kocaeli
  - Malatya
  - Sivas
- Ukraine (12):
  - Cherkasy
  - Chernivtsi
  - Dnipro
  - Ivano-Frankivsk
  - Kharkiv
  - Kiev
  - Kyiv
  - Lviv
  - Mykolayiv
  - Ternopil
  - Vinnytsia
  - Zaporizhzhya
- United Kingdom (11):
  - Llanelli, Carmarthenshire
  - Liverpool, Merseyside
  - Northampton, Northamptonshire
  - Carshalton, Surrey
  - Birmingham, West Midlands
  - Chichester, West Sussex
  - Bristol
  - Glasgow
  - London
  - Manchester
  - Middlesbrough
- Vietnam (2):
  - Hà Nội
  - Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, time point and process of data access. As such, Bayer commits to sharing upon request from qualified researcher's patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.

REFERENCES:
- [Result] Ruilope LM, Agarwal R, Anker SD, Bakris GL, Filippatos G, Nowack C, Kolkhof P, Joseph A, Mentenich N, Pitt B; FIGARO-DKD study investigators. Design and Baseline Characteristics of the Finerenone in Reducing Cardiovascular Mortality and Morbidity in Diabetic Kidney Disease Trial. Am J Nephrol. 2019;50(5):345-356. doi: 10.1159/000503712. Epub 2019 Oct 30. PMID 31665733
- [Result] Pitt B, Filippatos G, Agarwal R, Anker SD, Bakris GL, Rossing P, Joseph A, Kolkhof P, Nowack C, Schloemer P, Ruilope LM; FIGARO-DKD Investigators. Cardiovascular Events with Finerenone in Kidney Disease and Type 2 Diabetes. N Engl J Med. 2021 Dec 9;385(24):2252-2263. doi: 10.1056/NEJMoa2110956. Epub 2021 Aug 28. PMID 34449181
- [Derived] Mendoza JM, Weir MR, Anker SD, Filippatos G, Rossing P, Ahlers C, Brinker M, Fatoba ST, Horvat-Broecker A, Rohwedder K, Fornoni A; FIDELIO-DKD and FIGARO-DKD Investigators. Finerenone in People with CKD, Type 2 Diabetes, and History of Nephrectomy. Clin J Am Soc Nephrol. 2026 Jan 14. doi: 10.2215/CJN.0000000932. Online ahead of print. No abstract available. PMID 41533467
- [Derived] Katayama S, Anker SD, Zhu D, Kim S, Wu MJ, Kawanami D, Rossing P, Ruilope LM, Ahlers C, Brinker M, Mann A, Tian Y, Yamashita S, Pitt B; FIDELIO-DKD and FIGARO-DKD Investigators. Efficacy and safety of finerenone in Asian patients with type 2 diabetes and chronic kidney disease: A FIDELITY analysis by baseline kidney function. J Diabetes Complications. 2026 Jan;40(1):109213. doi: 10.1016/j.jdiacomp.2025.109213. Epub 2025 Nov 4. PMID 41289823
- [Derived] Ferreira JP, Mendonca L, Marques P, Neves JS, Zannad F, Packer M. Albuminuria Is the Key Driver of Kidney Benefit with Aldosterone Receptor Antagonists in Type 2 Diabetes. J Am Soc Nephrol. 2025 Sep 2. doi: 10.1681/ASN.0000000877. Online ahead of print. No abstract available. PMID 40892478
- [Derived] Rossing P, Birkenfeld AL, Fioretto P, McGill JB, Anker SD, Pitt B, Rohwedder K, Scalise A, Scott C, Filippatos G; FIDELIO-DKD and FIGARO-DKD Investigators. Finerenone and Clinical Outcomes in CKD and Type 2 Diabetes by Frailty Index: FIDELITY Post Hoc Analysis. Clin J Am Soc Nephrol. 2025 May 2;20(7):968-977. doi: 10.2215/CJN.0000000700. PMID 40315020
- [Derived] Singh AK, James G, Anker SD, Pitt B, Rossing P, Ruilope LM, Farjat AE, Farag YMK, Roberts L, Filippatos G; FIDELIO-DKD and FIGARO-DKD Investigators. Finerenone Efficacy in Patients with Chronic Kidney Disease, Type 2 Diabetes, and Anemia in FIDELITY. JACC Adv. 2025 Feb;4(2):101524. doi: 10.1016/j.jacadv.2024.101524. PMID 40021271
- [Derived] Pitt B, Agarwal R, Anker SD, Rossing P, Ruilope L, Herzog CA, Greenberg B, Pecoits-Filho R, Lambelet M, Lawatscheck R, Scalise A, Filippatos G. Hypokalaemia in patients with type 2 diabetes and chronic kidney disease: the effect of finerenone-a FIDELITY analysis. Eur Heart J Cardiovasc Pharmacother. 2025 Feb 8;11(1):10-19. doi: 10.1093/ehjcvp/pvae074. PMID 39380152
- [Derived] Bansal S, Canziani MEF, Birne R, Anker SD, Bakris GL, Filippatos G, Rossing P, Ruilope LM, Farjat AE, Kolkhof P, Lage A, Brinker M, Pitt B. Finerenone cardiovascular and kidney outcomes by age and sex: FIDELITY post hoc analysis of two phase 3, multicentre, double-blind trials. BMJ Open. 2024 Mar 19;14(3):e076444. doi: 10.1136/bmjopen-2023-076444. PMID 38508632
- [Derived] Agarwal R, Tu W, Farjat AE, Farag YMK, Toto R, Kaul S, Lawatscheck R, Rohwedder K, Ruilope LM, Rossing P, Pitt B, Filippatos G, Anker SD, Bakris GL; FIDELIO-DKD and FIGARO-DKD Investigators. Impact of Finerenone-Induced Albuminuria Reduction on Chronic Kidney Disease Outcomes in Type 2 Diabetes : A Mediation Analysis. Ann Intern Med. 2023 Dec;176(12):1606-1616. doi: 10.7326/M23-1023. Epub 2023 Dec 5. PMID 38048573
- [Derived] Flack JM, Agarwal R, Anker SD, Pitt B, Ruilope LM, Rossing P, Adler SG, Fried L, Jamerson K, Toto R, Brinker M, Farjat AE, Kolkhof P, Lawatscheck R, Joseph A, Bakris GL; FIDELIO-DKD and FIGARO-DKD Investigators. Finerenone in Black Patients With Type 2 Diabetes and CKD: A Post hoc Analysis of the Pooled FIDELIO-DKD and FIGARO-DKD Trials. Kidney Med. 2023 Sep 28;5(12):100730. doi: 10.1016/j.xkme.2023.100730. eCollection 2023 Dec. PMID 38046911
- [Derived] Rosas SE, Ruilope LM, Anker SD, Pitt B, Rossing P, Bonfanti AAC, Correa-Rotter R, Gonzalez F, Munoz CFJ, Pergola P, Umpierrez GE, Scalise A, Scott C, Lawatscheck R, Joseph A, Bakris GL; FIDELIO-DKD and FIGARO-DKD investigators. Finerenone in Hispanic Patients With CKD and Type 2 Diabetes: A Post Hoc FIDELITY Analysis. Kidney Med. 2023 Aug 1;5(10):100704. doi: 10.1016/j.xkme.2023.100704. eCollection 2023 Oct. PMID 37745646
- [Derived] Sarafidis P, Agarwal R, Pitt B, Wanner C, Filippatos G, Boletis J, Tuttle KR, Ruilope LM, Rossing P, Toto R, Anker SD, Liu ZH, Joseph A, Ahlers C, Brinker M, Lawatscheck R, Bakris G; FIDELIO-DKD and FIGARO-DKD Investigators. Outcomes with Finerenone in Participants with Stage 4 CKD and Type 2 Diabetes: A FIDELITY Subgroup Analysis. Clin J Am Soc Nephrol. 2023 May 1;18(5):602-612. doi: 10.2215/CJN.0000000000000149. Epub 2023 Apr 7. PMID 36927680
- [Derived] Agarwal R, Pitt B, Palmer BF, Kovesdy CP, Burgess E, Filippatos G, Malyszko J, Ruilope LM, Rossignol P, Rossing P, Pecoits-Filho R, Anker SD, Joseph A, Lawatscheck R, Wilson D, Gebel M, Bakris GL. A comparative post hoc analysis of finerenone and spironolactone in resistant hypertension in moderate-to-advanced chronic kidney disease. Clin Kidney J. 2022 Oct 30;16(2):293-302. doi: 10.1093/ckj/sfac234. eCollection 2023 Feb. PMID 36864892
- [Derived] Filippatos G, Anker SD, August P, Coats AJS, Januzzi JL, Mankovsky B, Rossing P, Ruilope LM, Pitt B, Sarafidis P, Teerlink JR, Kapelios CJ, Gebel M, Brinker M, Joseph A, Lage A, Bakris G, Agarwal R. Finerenone and effects on mortality in chronic kidney disease and type 2 diabetes: a FIDELITY analysis. Eur Heart J Cardiovasc Pharmacother. 2023 Feb 2;9(2):183-191. doi: 10.1093/ehjcvp/pvad001. PMID 36639130
- [Derived] Filippatos G, Anker SD, Pitt B, Rossing P, Joseph A, Kolkhof P, Lambelet M, Lawatscheck R, Bakris GL, Ruilope LM, Agarwal R. Finerenone and Heart Failure Outcomes by Kidney Function/Albuminuria in Chronic Kidney Disease and Diabetes. JACC Heart Fail. 2022 Nov;10(11):860-870. doi: 10.1016/j.jchf.2022.07.013. Epub 2022 Oct 12. PMID 36328655
- [Derived] Pitt B, Agarwal R, Anker SD, Ruilope LM, Rossing P, Ahlers C, Brinker M, Joseph A, Lambelet M, Lawatscheck R, Filippatos GS; FIDELIO-DKD and FIGARO-DKD Investigators. Association of Finerenone Use With Reduction in Treatment-Emergent Pneumonia and COVID-19 Adverse Events Among Patients With Type 2 Diabetes and Chronic Kidney Disease: A FIDELITY Pooled Secondary Analysis. JAMA Netw Open. 2022 Oct 3;5(10):e2236123. doi: 10.1001/jamanetworkopen.2022.36123. PMID 36287567
- [Derived] Filippatos G, Anker SD, Pitt B, McGuire DK, Rossing P, Ruilope LM, Butler J, Jankowska EA, Michos ED, Farmakis D, Farjat AE, Kolkhof P, Scalise A, Joseph A, Bakris GL, Agarwal R. Finerenone efficacy in patients with chronic kidney disease, type 2 diabetes and atherosclerotic cardiovascular disease. Eur Heart J Cardiovasc Pharmacother. 2022 Dec 15;9(1):85-93. doi: 10.1093/ehjcvp/pvac054. PMID 36251465
- [Derived] Filippatos G, Anker SD, Agarwal R, Ruilope LM, Rossing P, Bakris GL, Tasto C, Joseph A, Kolkhof P, Lage A, Pitt B; FIGARO-DKD Investigators. Finerenone Reduces Risk of Incident Heart Failure in Patients With Chronic Kidney Disease and Type 2 Diabetes: Analyses From the FIGARO-DKD Trial. Circulation. 2022 Feb 8;145(6):437-447. doi: 10.1161/CIRCULATIONAHA.121.057983. Epub 2021 Nov 13. PMID 34775784
- [Derived] Erraez S, Lopez-Mesa M, Gomez-Fernandez P. Mineralcorticoid receptor blockers in chronic kidney disease. Nefrologia (Engl Ed). 2021 May-Jun;41(3):258-275. doi: 10.1016/j.nefro.2020.10.001. Epub 2020 Dec 24. English, Spanish. PMID 33358451
- [Derived] Agarwal R, Anker SD, Bakris G, Filippatos G, Pitt B, Rossing P, Ruilope L, Gebel M, Kolkhof P, Nowack C, Joseph A; FIDELIO-DKD and FIGARO-DKD Investigators. Investigating new treatment opportunities for patients with chronic kidney disease in type 2 diabetes: the role of finerenone. Nephrol Dial Transplant. 2022 May 25;37(6):1014-1023. doi: 10.1093/ndt/gfaa294. PMID 33280027
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe. — http://www.clinicaltrialsregister.eu/
- See also: Click here to find results for studies related to Bayer products — http://clinicaltrials.bayer.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted at multiple centers in 48 countries/regions between 17-Sep-2015 (first participant first visit) and 02-Feb-2021 (last participant last visit).
Pre-assignment Details: Overall, 19381 participants were screened. Of them,11944 participants were screening failures and 7437 participants were randomized. 85 participants were prospectively excluded from the analyses due to critical GCP violations resulting in 7352 in full analysis set. 7341 participants received study treatment. 1 participant was assigned to placebo but received finerenone.
Groups:
- Finerenone: Participants received finerenone 10 mg or 20 mg once daily in addition to standard of care therapy
- Placebo: Participants received matching placebo once daily in addition to standard of care therapy
Period: Overall Study
Arm/Group | Finerenone | Placebo
Started (Randomized) | 3723 | 3714
Treated (One partcipant was randomized to placebo but received finerenone.) | 3683 | 3658
Included in FAS (85 participants were prospectively excluded from the analyses because of critical GCP violations) | 3686 | 3666
Completed (Participants (except those with critical GCP violations) were followed up regardless of having started treatment or not, and study completion is independent of administration of study treatment. A participant included in the FAS was considered as having completed the study if there was a contact with the participant after the end-of-study (EOS) notification or if the participant died.) | 3681 | 3653
Not Completed | 42 | 61
Not completed — Withdrawal by Subject | 1 | 7
Not completed — Lost to Follow-up | 4 | 6
Not completed — GCP violations | 37 | 48

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS): the FAS comprised all randomized participants (except those with critical GCP violations).
Groups:
- Total: Total of all reporting groups
Arm/Group | Finerenone | Placebo | Total
Number analyzed (Participants) | 3686 | 3666 | 7352
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.13 (9.67) | 64.13 (10.00) | 64.13 (9.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1158 | 1089 | 2247
  Male | 2528 | 2577 | 5105
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 618 | 603 | 1221
  Not Hispanic or Latino | 3058 | 3057 | 6115
  Unknown or Not Reported | 10 | 6 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 73 | 70 | 143
  Asian | 715 | 739 | 1454
  Native Hawaiian or Other Pacific Islander | 17 | 14 | 31
  Black or African American | 113 | 145 | 258
  White | 2672 | 2605 | 5277
  More than one race | 87 | 86 | 173
  Unknown or Not Reported | 9 | 7 | 16
Urinary albumin-to-creatinine ratio (UACR) [Median (Inter-Quartile Range); unit: milligram/gram (mg/g)] — Population: Participants in FAS with evaluable data
  milligram/gram (mg/g)
    number analyzed (Participants) | 3686 | 3664 | 7350
    (all) | 302.36 [105.47 to 749.05] | 315.06 [111.24 to 731.01] | 308.18 [108.09 to 739.86]
Estimated glomerular filtration rate (eGFR) [Mean (Standard Deviation); unit: mL/min/1.73m^2] — Population: Participants in FAS with evaluable data
  mL/min/1.73m^2
    number analyzed (Participants) | 3686 | 3665 | 7351
    (all) | 67.62 (21.65) | 67.99 (21.74) | 67.80 (21.69)

OUTCOME MEASURES:

1. Primary Outcome: The First Occurrence of the Composite Endpoint of Cardiovascular Death, Non-fatal Myocardial Infarction, Non Fatal Stroke, or Hospitalization for Heart Failure.
Description: Number of participants with the first occurrence of the primary cardiovascular (CV) composite outcome, CV death, non-fatal myocardial infarction (MI), non-fatal stroke, or hospitalization for heart failure were reported as descriptive result.
Time Frame: From randomization up until the first occurrence of the CV composite endpoint, or censoring at the end of the study, with an average study duration of 41 months.
Population: Full analysis set (FAS)
Measure: Count of Participants; unit: Participants
Arm/Group | Finerenone | Placebo
Number analyzed (Participants) | 3686 | 3666
Participants | 458 | 519
Statistical Analysis 1: Comparison: Finerenone vs Placebo; Test type: Superiority; p = 0.0264, Log Rank — A hierarchical testing procedure was used for the primary and secondary efficacy endpoints with each variable being tested at the adjusted two-sided significance level of 0.04967388; Stratified log rank test; Hazard Ratio (HR) = 0.87, 95% CI 2-sided [0.76 to 0.98] — A stratified Cox proportional hazards regression model was used to provide a point estimate of the hazard ratio and a corresponding two-sided 95% confidence interval

2. Secondary Outcome: The First Occurrence of the Composite Endpoint of Onset of Kidney Failure, a Sustained Decrease of eGFR ≥40% From Baseline Over at Least 4 Weeks, or Renal Death.
Description: Number of participants with first occurrence of the composite endpoint of onset of kidney failure, a sustained decrease of eGFR ≥40% from baseline over at least 4 weeks, or renal death were reported as descriptive result.
Time Frame: From randomization up until the first occurrence of the renal composite endpoint, or censoring at the end of the study, with an average study duration of 41 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Finerenone | Placebo
Number analyzed (Participants) | 3686 | 3666
Participants | 350 | 395
Statistical Analysis 1: Comparison: Finerenone vs Placebo; Test type: Superiority — If the treatment effect of the 40% renal composite endpoint was not significant, all other endpoints (i.e. all-cause hospitalization, all-cause mortality, change in UACR from baseline to Month 4, and 57% renal composite endpoint) would be tested in an exploratory manner; p = 0.0689, Log Rank — [p-value comment as in outcome 1, analysis 1]; Stratified log rank test; Hazard Ratio (HR) = 0.87, 95% CI 2-sided [0.76 to 1.01] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: All-cause Hospitalization
Description: Number of participants with first occurrence of a hospitalization event were reported as descriptive result.
Time Frame: From randomization up until the first occurrence of the hospitalization due to any cause, or censoring at the end of study, with an average study duration of 41 months
Population: Full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Finerenone | Placebo
Number analyzed (Participants) | 3686 | 3666
Participants | 1573 | 1605
Statistical Analysis 1: Comparison: Finerenone vs Placebo; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.3558, Log Rank — [p-value comment as in outcome 1, analysis 1]; Stratified log rank test; Hazard Ratio (HR) = 0.97, 95% CI 2-sided [0.90 to 1.04] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: All-cause Mortality
Description: Number of participants with death due to any cause were reported as descriptive result. Number of participants with outcome death reported here includes deaths occurred after randomization until the end of the study visit. Deaths after end of study visit are not included in this table.
Time Frame: From randomization up until death due to any cause, or censoring at the end of the study, with an average study duration of 41 months
Population: Full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Finerenone | Placebo
Number analyzed (Participants) | 3686 | 3666
Participants | 333 | 370
Statistical Analysis 1: Comparison: Finerenone vs Placebo; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.1337, Log Rank — [p-value comment as in outcome 1, analysis 1]; Stratified log rank test; Hazard Ratio (HR) = 0.89, 95% CI 2-sided [0.77 to 1.04] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Change in Urinary Albumin-to-creatine Ratio (UCAR) From Baseline to Month 4
Description: First morning void urine samples were collected to evaluate the urinary albumin-to-creatinine ratio (UACR). Month 4 was the visit closest to day 120 within a time window of 120 ± 30 days after randomization. If no measurements were available in this time window, the participant was excluded from this analysis. Ratio of UACR at Month 4 to UACR at baseline is reported as the change.
Time Frame: From baseline up until Month 4
Population: Subjects in full analysis set with measurements available within the time window of Month 4
Measure: Least Squares Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Finerenone | Placebo
Number analyzed (Participants) | 3521 | 3476
Ratio | 0.624 [0.606 to 0.642] | 0.922 [0.896 to 0.949]
Statistical Analysis 1: Comparison: Finerenone vs Placebo; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p < 0.0001, ANCOVA — P-value from F-test of equal means between the treatment groups. A hierarchical testing procedure was used for the primary and secondary efficacy endpoints with each variable being tested at the adjusted two-sided significance level of 0.04967388; Ratio of least squares means = 0.676, 95% CI 2-sided [0.650 to 0.704]

6. Secondary Outcome: The First Occurrence of the Composite Endpoint of Onset of Kidney Failure, a Sustained Decrease in eGFR of ≥57% From Baseline Over at Least 4 Weeks, or Renal Death
Description: Number of participants with first occurrence of the renal composite outcome, onset of kidney failure, a sustained decrease in eGFR of ≥57% from baseline over at least 4 weeks, or renal death were reported as descriptive result.
Time Frame: as for outcome 2
Population: Full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Finerenone | Placebo
Number analyzed (Participants) | 3686 | 3666
Participants | 108 | 139
Statistical Analysis 1: Comparison: Finerenone vs Placebo; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.0406, Log Rank — [p-value comment as in outcome 1, analysis 1]; Stratified log rank test; Hazard Ratio (HR) = 0.77, 95% CI 2-sided [0.60 to 0.99] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: After the first dose of study drug up to 3 days after any temporary or permanent interruption of study drug, with an average treatment duration of 36 months.
Description: Adverse events are reported for the safety analysis set (SAF) that comprised all randomized participants who took at least 1 dose of study drug (except those with critical GCP violations). Adverse events for all-cause mortality are reported for the Full analysis set (FAS) that comprised all randomized participants (except those with critical GCP violations) and considers all deaths after randomization, including those after the end of study visit.
Arm/Group | Finerenone | Placebo
All-Cause Mortality (participants affected / at risk) | 339/3686 | 383/3666
Serious Adverse Events (participants affected / at risk) | 1158/3683 | 1215/3658
Other Adverse Events (participants affected / at risk) | 1797/3683 | 1717/3658
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Finerenone (N=3683) | Placebo (N=3658)
Anaemia (Blood and lymphatic system disorders) | 18 (21) | 15 (15)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hilar lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hypocoagulable state (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Lymphadenopathy mediastinal (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Microcytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hypereosinophilic syndrome (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acquired haemophilia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Bicytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Blood loss anaemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 2 (2)
Angina pectoris (Cardiac disorders) | 2 (2) | 2 (2)
Angina unstable (Cardiac disorders) | 4 (4) | 1 (1)
Aortic valve disease mixed (Cardiac disorders) | 2 (2) | 0 (0)
Aortic valve incompetence (Cardiac disorders) | 0 (0) | 1 (1)
Aortic valve stenosis (Cardiac disorders) | 3 (3) | 3 (4)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 4 (4) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 2 (2)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 2 (2)
Atrioventricular block second degree (Cardiac disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 3 (3) | 2 (2)
Bundle branch block left (Cardiac disorders) | 0 (0) | 2 (2)
Cardiac arrest (Cardiac disorders) | 1 (1) | 2 (2)
Cardiac failure (Cardiac disorders) | 5 (5) | 10 (10)
Cardiac failure acute (Cardiac disorders) | 4 (4) | 0 (0)
Cardiac failure chronic (Cardiac disorders) | 2 (2) | 3 (4)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Cor pulmonale chronic (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 5 (5) | 6 (6)
Coronary artery occlusion (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 2 (2) | 2 (2)
Extrasystoles (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 3 (3) | 3 (3)
Palpitations (Cardiac disorders) | 1 (1) | 1 (1)
Pericardial haemorrhage (Cardiac disorders) | 1 (1) | 0 (0)
Pericarditis (Cardiac disorders) | 2 (2) | 0 (0)
Sinoatrial block (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 2 (2) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Left ventricular hypertrophy (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular hypokinesia (Cardiac disorders) | 1 (1) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 1 (1)
Pulseless electrical activity (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac valve disease (Cardiac disorders) | 0 (0) | 1 (1)
Acute left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular tachyarrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Sinus node dysfunction (Cardiac disorders) | 1 (1) | 2 (2)
Paroxysmal atrioventricular block (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Arnold-Chiari malformation (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Hypospadias (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Phimosis (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Adenomatous polyposis coli (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Anomaly of middle ear congenital (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Deafness (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Tympanic membrane perforation (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 7 (7) | 6 (6)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Vestibular ataxia (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vestibular disorder (Ear and labyrinth disorders) | 0 (0) | 2 (2)
Sudden hearing loss (Ear and labyrinth disorders) | 2 (2) | 3 (3)
Acute vestibular syndrome (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Goitre (Endocrine disorders) | 2 (2) | 0 (0)
Hyperparathyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Primary hyperaldosteronism (Endocrine disorders) | 1 (1) | 0 (0)
Toxic nodular goitre (Endocrine disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 15 (18) | 11 (16)
Cataract diabetic (Eye disorders) | 1 (2) | 1 (1)
Cataract nuclear (Eye disorders) | 0 (0) | 2 (2)
Dermatochalasis (Eye disorders) | 0 (0) | 1 (1)
Diabetic eye disease (Eye disorders) | 1 (1) | 0 (0)
Diabetic retinopathy (Eye disorders) | 11 (21) | 7 (8)
Diplopia (Eye disorders) | 1 (1) | 0 (0)
Extraocular muscle paresis (Eye disorders) | 1 (1) | 0 (0)
Eye haemorrhage (Eye disorders) | 2 (2) | 1 (1)
Glaucoma (Eye disorders) | 4 (4) | 3 (3)
Macular oedema (Eye disorders) | 1 (12) | 3 (4)
Ophthalmoplegia (Eye disorders) | 0 (0) | 1 (1)
Optic ischaemic neuropathy (Eye disorders) | 0 (0) | 1 (1)
Retinal detachment (Eye disorders) | 2 (2) | 3 (3)
Retinal haemorrhage (Eye disorders) | 1 (1) | 3 (4)
Retinopathy (Eye disorders) | 1 (1) | 0 (0)
Retinopathy proliferative (Eye disorders) | 1 (1) | 1 (1)
Vision blurred (Eye disorders) | 1 (1) | 0 (0)
Vitreous haemorrhage (Eye disorders) | 16 (23) | 7 (8)
Macular hole (Eye disorders) | 0 (0) | 2 (2)
Eyelid cyst (Eye disorders) | 0 (0) | 1 (1)
Age-related macular degeneration (Eye disorders) | 1 (1) | 0 (0)
Ulcerative keratitis (Eye disorders) | 1 (1) | 0 (0)
Rhegmatogenous retinal detachment (Eye disorders) | 1 (1) | 0 (0)
Ocular ischaemic syndrome (Eye disorders) | 1 (1) | 0 (0)
Macular fibrosis (Eye disorders) | 3 (3) | 2 (3)
Abdominal adhesions (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal mass (Gastrointestinal disorders) | 0 (0) | 1 (2)
Abdominal pain (Gastrointestinal disorders) | 5 (5) | 6 (6)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 4 (4) | 4 (4)
Anal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 3 (3)
Barrett's oesophagus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chronic gastritis (Gastrointestinal disorders) | 2 (2) | 2 (2)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 2 (2) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 7 (8) | 4 (4)
Diverticulum (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 3 (3) | 2 (2)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 1 (2)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastric haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastric polyps (Gastrointestinal disorders) | 0 (0) | 2 (3)
Gastric ulcer (Gastrointestinal disorders) | 2 (2) | 1 (1)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 2 (2)
Gastritis (Gastrointestinal disorders) | 2 (2) | 2 (2)
Gastritis erosive (Gastrointestinal disorders) | 1 (1) | 2 (2)
Gastritis haemorrhagic (Gastrointestinal disorders) | 2 (2) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 4 (4)
Gastroduodenal ulcer (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 7 (7) | 9 (12)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Haemorrhoids (Gastrointestinal disorders) | 4 (4) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus paralytic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Impaired gastric emptying (Gastrointestinal disorders) | 0 (0) | 2 (2)
Inguinal hernia (Gastrointestinal disorders) | 2 (2) | 9 (10)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 7 (11)
Melaena (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mesenteric vein thrombosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mouth haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Oesophageal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatic cyst (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 5 (7) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 12 (16) | 4 (4)
Pancreatitis chronic (Gastrointestinal disorders) | 2 (2) | 3 (3)
Pancreatitis necrotising (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis relapsing (Gastrointestinal disorders) | 0 (0) | 1 (1)
Parotid gland enlargement (Gastrointestinal disorders) | 1 (1) | 0 (0)
Peptic ulcer (Gastrointestinal disorders) | 2 (2) | 0 (0)
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 3 (3) | 3 (4)
Rectal polyp (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (4) | 4 (4)
Small intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Swollen tongue (Gastrointestinal disorders) | 1 (1) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 1 (1) | 2 (2)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 4 (4) | 6 (6)
Volvulus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 5 (5) | 3 (3)
Pancreatic mass (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal discharge (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anal haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastric dysplasia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal dysplasia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Subileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Mechanical ileus (Gastrointestinal disorders) | 2 (2) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 14 (16) | 11 (13)
Oesophageal polyp (Gastrointestinal disorders) | 0 (0) | 1 (1)
Internal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oedematous pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Varices oesophageal (Gastrointestinal disorders) | 1 (6) | 0 (0)
Gastric varices haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Reflux gastritis (Gastrointestinal disorders) | 0 (0) | 1 (2)
Gastrointestinal oedema (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal mass (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal symptom (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric mucosal lesion (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diverticular perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Salivary gland disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Incarcerated umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatic duct stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal wall haematoma (Gastrointestinal disorders) | 0 (0) | 2 (2)
Haemorrhagic erosive gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal wall haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Omental infarction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Functional gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal hernia perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dental cyst (Gastrointestinal disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 3 (3) | 2 (2)
Chest pain (General disorders) | 18 (18) | 20 (22)
Death (General disorders) | 8 (8) | 6 (6)
Generalised oedema (General disorders) | 0 (0) | 1 (1)
Impaired healing (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 3 (3)
Oedema (General disorders) | 2 (2) | 2 (2)
Oedema peripheral (General disorders) | 1 (1) | 9 (21)
Pain (General disorders) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 6 (6) | 5 (6)
Sudden death (General disorders) | 0 (0) | 1 (1)
Peripheral swelling (General disorders) | 2 (2) | 1 (1)
General physical health deterioration (General disorders) | 2 (2) | 8 (10)
Oedema due to cardiac disease (General disorders) | 1 (1) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 1 (1) | 1 (1)
Haemorrhagic cyst (General disorders) | 0 (0) | 1 (1)
Adhesion (General disorders) | 0 (0) | 1 (1)
Polyp (General disorders) | 1 (1) | 1 (1)
Drug intolerance (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 3 (4)
Complication associated with device (General disorders) | 1 (1) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 2 (2) | 2 (2)
Hanging (General disorders) | 1 (1) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 5 (5) | 3 (5)
Biliary colic (Hepatobiliary disorders) | 2 (2) | 1 (2)
Biliary fistula (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 2 (2) | 3 (3)
Cholangitis acute (Hepatobiliary disorders) | 1 (1) | 2 (2)
Cholecystitis (Hepatobiliary disorders) | 7 (7) | 5 (5)
Cholecystitis acute (Hepatobiliary disorders) | 9 (10) | 7 (7)
Cholecystitis chronic (Hepatobiliary disorders) | 3 (3) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 5 (5) | 7 (9)
Chronic hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cirrhosis alcoholic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Fatty liver alcoholic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1) | 2 (2)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatorenal syndrome (Hepatobiliary disorders) | 1 (1) | 0 (0)
Jaundice (Hepatobiliary disorders) | 0 (0) | 1 (1)
Jaundice cholestatic (Hepatobiliary disorders) | 1 (1) | 2 (2)
Liver disorder (Hepatobiliary disorders) | 1 (1) | 0 (0)
Portal hypertension (Hepatobiliary disorders) | 0 (0) | 1 (3)
Portal vein thrombosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystocholangitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Gallbladder polyp (Hepatobiliary disorders) | 0 (0) | 1 (1)
Non-alcoholic steatohepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Biliary dyskinesia (Hepatobiliary disorders) | 2 (2) | 0 (0)
Primary biliary cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1)
Anaphylactic shock (Immune system disorders) | 1 (1) | 1 (1)
Abdominal wall abscess (Infections and infestations) | 1 (1) | 0 (0)
Abscess (Infections and infestations) | 0 (0) | 2 (2)
Acute sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Anorectal cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 5 (5) | 5 (5)
Arteriosclerotic gangrene (Infections and infestations) | 0 (0) | 1 (1)
Aspergilloma (Infections and infestations) | 2 (2) | 0 (0)
Atypical pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 2 (2) | 0 (0)
Bronchitis (Infections and infestations) | 7 (7) | 9 (9)
Campylobacter gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 40 (46) | 28 (29)
Cellulitis gangrenous (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis staphylococcal (Infections and infestations) | 0 (0) | 1 (1)
Chronic hepatitis C (Infections and infestations) | 0 (0) | 1 (1)
Chronic sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Corneal abscess (Infections and infestations) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 4 (4) | 4 (4)
Dengue fever (Infections and infestations) | 1 (1) | 0 (0)
Diabetic gangrene (Infections and infestations) | 1 (1) | 1 (1)
Diverticulitis (Infections and infestations) | 4 (4) | 4 (4)
Diverticulitis intestinal haemorrhagic (Infections and infestations) | 1 (1) | 0 (0)
Endocarditis (Infections and infestations) | 1 (1) | 0 (0)
Enterococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Epididymitis (Infections and infestations) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 10 (12) | 15 (21)
Escherichia sepsis (Infections and infestations) | 0 (0) | 1 (1)
Eye infection (Infections and infestations) | 0 (0) | 1 (1)
Fournier's gangrene (Infections and infestations) | 0 (0) | 1 (1)
Furuncle (Infections and infestations) | 0 (0) | 1 (1)
Gangrene (Infections and infestations) | 5 (5) | 6 (7)
Gastroenteritis (Infections and infestations) | 11 (12) | 15 (15)
Gastroenteritis rotavirus (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis salmonella (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 3 (3) | 0 (0)
Herpes zoster (Infections and infestations) | 3 (3) | 1 (1)
HIV infection (Infections and infestations) | 1 (1) | 0 (0)
Infected skin ulcer (Infections and infestations) | 2 (2) | 1 (1)
Infection (Infections and infestations) | 1 (1) | 5 (5)
Infectious mononucleosis (Infections and infestations) | 1 (1) | 0 (0)
Infective myositis (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 5 (5) | 6 (6)
Labyrinthitis (Infections and infestations) | 0 (0) | 2 (2)
Localised infection (Infections and infestations) | 9 (10) | 6 (6)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 5 (5)
Mastoiditis (Infections and infestations) | 1 (1) | 0 (0)
Meningitis (Infections and infestations) | 1 (1) | 0 (0)
Necrotising fasciitis (Infections and infestations) | 1 (1) | 2 (2)
Orchitis (Infections and infestations) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 12 (16) | 13 (13)
Osteomyelitis acute (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis chronic (Infections and infestations) | 3 (3) | 2 (2)
Otitis externa (Infections and infestations) | 2 (2) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 1 (1)
Paronychia (Infections and infestations) | 0 (0) | 1 (1)
Pelvic inflammatory disease (Infections and infestations) | 0 (0) | 1 (1)
Peritonitis (Infections and infestations) | 1 (1) | 0 (0)
Peritonsillar abscess (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Pilonidal cyst (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 73 (77) | 113 (121)
Pneumonia haemophilus (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia influenzal (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia klebsiella (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia legionella (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia pneumococcal (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia streptococcal (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia viral (Infections and infestations) | 2 (2) | 1 (1)
Postoperative wound infection (Infections and infestations) | 7 (7) | 2 (2)
Prostatic abscess (Infections and infestations) | 1 (1) | 0 (0)
Pulmonary mycosis (Infections and infestations) | 1 (1) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 1 (1) | 2 (2)
Pyelitis (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 9 (9) | 4 (4)
Pyelonephritis acute (Infections and infestations) | 4 (4) | 2 (2)
Pyelonephritis chronic (Infections and infestations) | 1 (1) | 2 (2)
Salpingitis (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 16 (16) | 20 (21)
Septic shock (Infections and infestations) | 4 (4) | 5 (5)
Sialoadenitis (Infections and infestations) | 1 (2) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 4 (4)
Subacute endocarditis (Infections and infestations) | 0 (0) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 4 (4) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 1 (1)
Tracheobronchitis (Infections and infestations) | 0 (0) | 1 (1)
Tuberculosis (Infections and infestations) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 5 (5)
Urinary tract infection (Infections and infestations) | 28 (33) | 39 (40)
Vestibular neuronitis (Infections and infestations) | 0 (0) | 2 (2)
Viral infection (Infections and infestations) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 2 (2) | 4 (4)
Urosepsis (Infections and infestations) | 12 (15) | 13 (13)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1)
Anal abscess (Infections and infestations) | 2 (2) | 4 (4)
Sinobronchitis (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection fungal (Infections and infestations) | 1 (1) | 0 (0)
Abscess limb (Infections and infestations) | 9 (12) | 5 (5)
Abscess soft tissue (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Pulmonary sepsis (Infections and infestations) | 0 (0) | 2 (2)
Gastritis viral (Infections and infestations) | 0 (0) | 1 (1)
Coronavirus infection (Infections and infestations) | 0 (0) | 1 (1)
Febrile infection (Infections and infestations) | 1 (1) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Perirectal abscess (Infections and infestations) | 0 (0) | 1 (1)
Arthritis bacterial (Infections and infestations) | 1 (1) | 1 (1)
Abscess neck (Infections and infestations) | 1 (1) | 0 (0)
Bacterial sepsis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection bacterial (Infections and infestations) | 0 (0) | 1 (1)
Stenotrophomonas sepsis (Infections and infestations) | 0 (0) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 1 (1)
Escherichia bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 1 (1) | 1 (1)
Abdominal infection (Infections and infestations) | 1 (1) | 0 (0)
Catheter site infection (Infections and infestations) | 0 (0) | 1 (1)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 (1) | 3 (4)
Periorbital cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Infective tenosynovitis (Infections and infestations) | 1 (1) | 0 (0)
Abdominal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1)
Acute hepatitis B (Infections and infestations) | 0 (0) | 1 (1)
Intervertebral discitis (Infections and infestations) | 2 (2) | 2 (2)
Diabetic foot infection (Infections and infestations) | 7 (9) | 5 (6)
Bacterial infection (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 2 (2) | 7 (7)
Arthritis infective (Infections and infestations) | 1 (1) | 0 (0)
Genitourinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Tracheobronchitis viral (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis bacterial (Infections and infestations) | 2 (2) | 0 (0)
Soft tissue infection (Infections and infestations) | 1 (1) | 3 (3)
Respiratory tract infection (Infections and infestations) | 6 (6) | 4 (4)
Cholecystitis infective (Infections and infestations) | 1 (1) | 2 (2)
Device related infection (Infections and infestations) | 0 (0) | 1 (1)
Otitis externa bacterial (Infections and infestations) | 1 (1) | 0 (0)
Cystitis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Enterocolitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Lymphadenitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Wound infection bacterial (Infections and infestations) | 1 (1) | 0 (0)
Post procedural infection (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis norovirus (Infections and infestations) | 1 (1) | 1 (1)
Emphysematous pyelonephritis (Infections and infestations) | 2 (2) | 0 (0)
Gastrointestinal viral infection (Infections and infestations) | 0 (0) | 1 (1)
Infective exacerbation of bronchiectasis (Infections and infestations) | 0 (0) | 2 (2)
Infectious pleural effusion (Infections and infestations) | 1 (1) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster meningoencephalitis (Infections and infestations) | 0 (0) | 1 (1)
Medical device site infection (Infections and infestations) | 1 (1) | 0 (0)
Intestinal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Spinal cord abscess (Infections and infestations) | 1 (1) | 0 (0)
Necrotising soft tissue infection (Infections and infestations) | 1 (1) | 0 (0)
Infected bite (Infections and infestations) | 0 (0) | 1 (1)
Vascular device infection (Infections and infestations) | 0 (0) | 1 (1)
Large intestine infection (Infections and infestations) | 0 (0) | 2 (2)
Vascular graft infection (Infections and infestations) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 17 (17) | 22 (22)
COVID-19 pneumonia (Infections and infestations) | 9 (9) | 11 (11)
Accident (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Acetabulum fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 6 (6) | 6 (6)
Cartilage injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cystitis radiation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 4 (4) | 5 (5)
Femoral neck fracture (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 8 (8) | 8 (8)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
Foreign body aspiration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gun shot wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Hip fracture (Injury, poisoning and procedural complications) | 5 (6) | 2 (2)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 4 (4)
Injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Injury corneal (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Multiple fractures (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Multiple injuries (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Patella fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radiation proctitis (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 2 (2) | 5 (5)
Rib fracture (Injury, poisoning and procedural complications) | 4 (4) | 4 (4)
Road traffic accident (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Scapula fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Skull fractured base (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 2 (2) | 2 (3)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Splenic injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 3 (3) | 6 (6)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
Tendon rupture (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)
Tibia fracture (Injury, poisoning and procedural complications) | 5 (6) | 1 (1)
Traumatic ulcer (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ulna fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Anaemia postoperative (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Traumatic fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 4 (5) | 2 (2)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Brain contusion (Injury, poisoning and procedural complications) | 1 (2) | 2 (2)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Intervertebral disc injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cardiac procedure complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Abdominal injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
Poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skull fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Chest injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Upper limb fracture (Injury, poisoning and procedural complications) | 2 (3) | 0 (0)
Postoperative wound complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Stomal hernia (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular anastomosis aneurysm (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cerebral hyperperfusion syndrome (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Bone contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Heat illness (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Wound contamination (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Periprosthetic fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Craniocerebral injury (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skin wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Meniscus injury (Injury, poisoning and procedural complications) | 4 (4) | 2 (2)
Eye contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural intestinal perforation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Postoperative delirium (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Dental restoration failure (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ocular procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Reproductive tract procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Arthroscopy (Investigations) | 0 (0) | 3 (3)
Biopsy bladder (Investigations) | 1 (1) | 0 (0)
Biopsy kidney (Investigations) | 0 (0) | 1 (2)
Biopsy liver (Investigations) | 0 (0) | 1 (1)
Biopsy prostate (Investigations) | 0 (0) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 2 (2) | 3 (3)
Blood glucose increased (Investigations) | 4 (4) | 4 (4)
Blood magnesium decreased (Investigations) | 0 (0) | 1 (1)
Blood potassium decreased (Investigations) | 1 (1) | 0 (0)
Blood potassium increased (Investigations) | 2 (2) | 0 (0)
Blood pressure increased (Investigations) | 1 (1) | 2 (2)
C-reactive protein increased (Investigations) | 1 (2) | 1 (1)
Colonoscopy (Investigations) | 4 (4) | 2 (2)
Colonoscopy normal (Investigations) | 1 (1) | 0 (0)
Computerised tomogram (Investigations) | 1 (1) | 0 (0)
Electrocardiogram abnormal (Investigations) | 1 (1) | 1 (1)
Endoscopy (Investigations) | 2 (2) | 0 (0)
Glomerular filtration rate decreased (Investigations) | 4 (4) | 1 (1)
Glycosylated haemoglobin increased (Investigations) | 1 (1) | 3 (3)
Haematocrit decreased (Investigations) | 1 (1) | 0 (0)
Blood urine present (Investigations) | 0 (0) | 1 (1)
International normalised ratio increased (Investigations) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 1 (1)
Angiogram cerebral (Investigations) | 0 (0) | 1 (1)
Sleep study (Investigations) | 1 (1) | 0 (0)
Blood pressure orthostatic decreased (Investigations) | 1 (1) | 0 (0)
Troponin increased (Investigations) | 0 (0) | 1 (1)
Cardiac function test abnormal (Investigations) | 1 (1) | 0 (0)
Anticoagulation drug level below therapeutic (Investigations) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 0 (0) | 1 (1)
Angiogram (Investigations) | 1 (1) | 0 (0)
Investigation (Investigations) | 1 (1) | 0 (0)
Respiratory syncytial virus test positive (Investigations) | 0 (0) | 1 (1)
Influenza A virus test positive (Investigations) | 0 (0) | 4 (4)
Endobronchial ultrasound (Investigations) | 0 (0) | 1 (1)
Gastrointestinal stoma output increased (Investigations) | 0 (0) | 1 (1)
Liver function test increased (Investigations) | 0 (0) | 2 (2)
Cancer staging (Investigations) | 1 (1) | 0 (0)
Angiocardiogram (Investigations) | 1 (1) | 0 (0)
SARS-CoV-2 test positive (Investigations) | 0 (0) | 1 (1)
SARS-CoV-2 test negative (Investigations) | 0 (0) | 1 (1)
Cachexia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 8 (8) | 10 (10)
Diabetes mellitus (Metabolism and nutrition disorders) | 20 (24) | 25 (31)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 27 (34) | 17 (20)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 3 (3) | 8 (8)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Gout (Metabolism and nutrition disorders) | 2 (3) | 2 (2)
Hypercalcaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 23 (24) | 11 (11)
Hyperkalaemia (Metabolism and nutrition disorders) | 23 (25) | 4 (6)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 17 (20) | 28 (31)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 6 (7)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 6 (7) | 7 (9)
Hypovolaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Obesity (Metabolism and nutrition disorders) | 4 (4) | 3 (3)
Metabolic syndrome (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Metabolic disorder (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diabetic complication (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Mineral metabolism disorder (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 2 (2) | 3 (3)
Periarthritis calcarea (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 33 (45) | 25 (33)
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 18 (20) | 13 (16)
Ankylosing spondylitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (6) | 6 (7)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (2) | 3 (3)
Arthritis reactive (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (10) | 3 (3)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Chondromalacia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Exostosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Fasciitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (5)
Neuropathic arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Osteitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 22 (23) | 9 (11)
Osteolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Plantar fascial fibromatosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (13)
Resorption bone increased (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (4)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 4 (4) | 4 (4)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 8 (10) | 9 (9)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spondyloarthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Soft tissue haemorrhage (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Facet joint syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc compression (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tenosynovitis stenosans (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal ligament ossification (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Inclusion body myositis (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Diastasis recti abdominis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tendon discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Vertebral lateral recess stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Immobilisation syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (2)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 2 (2)
Adrenal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 4 (4)
Benign neoplasm of bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Benign neoplasm of prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 11 (13) | 4 (4)
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (4) | 0 (0)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 3 (3)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 3 (3)
Bone cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 4 (4)
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 14 (15) | 9 (10)
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Enchondromatosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Haemangioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hypergammaglobulinaemia benign monoclonal (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hypopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Laryngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 4 (4)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Meningioma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neoplasm prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 5 (5)
Oropharyngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 5 (5)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pituitary tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 1 (1)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3)
Respiratory papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Seminoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (3) | 2 (2)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma of the oral cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Thymoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (4) | 1 (2)
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Tumour ulceration (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Salivary gland adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colorectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gastrointestinal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ear neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Retroperitoneal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Choroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Testis cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (3)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (7) | 8 (8)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Pancreatic carcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 (10) | 24 (24)
Benign anorectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Benign gastrointestinal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Benign pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Female reproductive neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Anal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (3)
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (4) | 2 (3)
Ovarian neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Adrenal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Oesophageal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 5 (6)
Rectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tumour invasion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Bladder transitional cell carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Haemangioma of spleen (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Epithelioid mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 4 (4)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (4) | 2 (2)
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Invasive papillary breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Papillary cystadenoma lymphomatosum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Triple negative breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Invasive breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Transitional cell carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Papillary renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Squamous cell carcinoma of the parotid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Altered state of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Amnesia (Nervous system disorders) | 1 (1) | 0 (0)
Aphasia (Nervous system disorders) | 1 (1) | 1 (1)
Ataxia (Nervous system disorders) | 0 (0) | 1 (1)
Brain stem haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 3 (3) | 4 (4)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Cauda equina syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 3 (3) | 0 (0)
Cerebrospinal fluid leakage (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular disorder (Nervous system disorders) | 1 (1) | 2 (2)
Cervicobrachial syndrome (Nervous system disorders) | 1 (1) | 1 (1)
Coma (Nervous system disorders) | 0 (0) | 1 (1)
Dementia (Nervous system disorders) | 0 (0) | 1 (1)
Dementia Alzheimer's type (Nervous system disorders) | 1 (2) | 1 (1)
Diabetic hyperosmolar coma (Nervous system disorders) | 0 (0) | 1 (1)
Diabetic ketoacidotic hyperglycaemic coma (Nervous system disorders) | 0 (0) | 1 (1)
Diabetic neuropathy (Nervous system disorders) | 11 (13) | 7 (9)
Dizziness (Nervous system disorders) | 7 (10) | 8 (8)
Dizziness postural (Nervous system disorders) | 1 (1) | 1 (1)
Dysarthria (Nervous system disorders) | 1 (1) | 0 (0)
Dyskinesia (Nervous system disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 2 (2)
Epilepsy (Nervous system disorders) | 2 (3) | 1 (1)
Facial paralysis (Nervous system disorders) | 4 (5) | 2 (2)
Generalised tonic-clonic seizure (Nervous system disorders) | 1 (1) | 1 (1)
Guillain-Barre syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 0 (0)
Hemiparesis (Nervous system disorders) | 2 (2) | 1 (1)
Hepatic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1)
Hypertensive encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Hypoglycaemic coma (Nervous system disorders) | 0 (0) | 1 (1)
IIIrd nerve paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Intracranial aneurysm (Nervous system disorders) | 0 (0) | 1 (1)
Intraventricular haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 1 (1) | 1 (1)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0)
Meralgia paraesthetica (Nervous system disorders) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 1 (1)
Moyamoya disease (Nervous system disorders) | 1 (1) | 0 (0)
Myelopathy (Nervous system disorders) | 2 (2) | 1 (1)
Neuralgia (Nervous system disorders) | 1 (1) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1)
Normal pressure hydrocephalus (Nervous system disorders) | 3 (3) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Polyneuropathy (Nervous system disorders) | 1 (1) | 1 (1)
Presyncope (Nervous system disorders) | 3 (3) | 2 (2)
Radiculopathy (Nervous system disorders) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 3 (3) | 1 (1)
Seizure (Nervous system disorders) | 2 (2) | 1 (1)
Sensory disturbance (Nervous system disorders) | 1 (1) | 1 (2)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1)
Spinal cord compression (Nervous system disorders) | 1 (1) | 1 (1)
Spondylitic myelopathy (Nervous system disorders) | 0 (0) | 2 (2)
Subarachnoid haemorrhage (Nervous system disorders) | 4 (4) | 4 (4)
Syncope (Nervous system disorders) | 14 (14) | 16 (16)
Tension headache (Nervous system disorders) | 1 (1) | 0 (0)
Toxic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 2 (2) | 2 (2)
Ulnar neuritis (Nervous system disorders) | 1 (1) | 0 (0)
Vascular headache (Nervous system disorders) | 2 (3) | 0 (0)
Vertigo CNS origin (Nervous system disorders) | 0 (0) | 1 (1)
Balance disorder (Nervous system disorders) | 1 (1) | 1 (1)
Cervical radiculopathy (Nervous system disorders) | 0 (0) | 3 (5)
Lumbar radiculopathy (Nervous system disorders) | 1 (1) | 2 (2)
Dysstasia (Nervous system disorders) | 0 (0) | 1 (1)
Lacunar infarction (Nervous system disorders) | 1 (1) | 2 (2)
Facial paresis (Nervous system disorders) | 0 (0) | 3 (3)
Chronic inflammatory demyelinating polyradiculoneuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Cognitive disorder (Nervous system disorders) | 1 (1) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 2 (2) | 0 (0)
Partial seizures (Nervous system disorders) | 1 (1) | 0 (0)
Facial nerve disorder (Nervous system disorders) | 0 (0) | 1 (1)
Parkinson's disease (Nervous system disorders) | 0 (0) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 2 (2) | 0 (0)
Mononeuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Vascular encephalopathy (Nervous system disorders) | 2 (2) | 0 (0)
Hypoglycaemic unconsciousness (Nervous system disorders) | 1 (1) | 1 (1)
Amputation stump pain (Nervous system disorders) | 1 (1) | 0 (0)
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Hyperglycaemic unconsciousness (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral nerve paresis (Nervous system disorders) | 0 (0) | 1 (1)
Intensive care unit acquired weakness (Nervous system disorders) | 0 (0) | 1 (1)
Posthaemorrhagic hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1)
Central nervous system vasculitis (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (2) | 0 (0)
Completed suicide (Psychiatric disorders) | 2 (2) | 0 (0)
Confusional state (Psychiatric disorders) | 2 (2) | 1 (1)
Delusional disorder, unspecified type (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 2 (2) | 2 (2)
Drug abuse (Psychiatric disorders) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 2 (2) | 2 (2)
Bipolar disorder (Psychiatric disorders) | 1 (2) | 0 (0)
Major depression (Psychiatric disorders) | 1 (3) | 1 (1)
Mental disorder due to a general medical condition (Psychiatric disorders) | 1 (1) | 0 (0)
Suicide threat (Psychiatric disorders) | 0 (0) | 1 (1)
Albuminuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Azotaemia (Renal and urinary disorders) | 0 (0) | 1 (1)
Calculus bladder (Renal and urinary disorders) | 3 (4) | 1 (1)
Calculus urinary (Renal and urinary disorders) | 2 (2) | 3 (3)
Glomerulonephritis chronic (Renal and urinary disorders) | 0 (0) | 1 (1)
Glomerulonephritis membranous (Renal and urinary disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 5 (5) | 6 (6)
Hydronephrosis (Renal and urinary disorders) | 2 (2) | 4 (4)
Nephrolithiasis (Renal and urinary disorders) | 12 (13) | 8 (11)
Nephropathy (Renal and urinary disorders) | 2 (2) | 2 (2)
Nephrotic syndrome (Renal and urinary disorders) | 0 (0) | 2 (2)
Proteinuria (Renal and urinary disorders) | 0 (0) | 2 (2)
Renal artery stenosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal colic (Renal and urinary disorders) | 3 (4) | 2 (2)
Renal cyst (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 4 (4) | 2 (2)
Ureteric obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary hesitation (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 2 (2) | 0 (0)
Urinary retention (Renal and urinary disorders) | 5 (5) | 5 (5)
Urinary tract disorder (Renal and urinary disorders) | 0 (0) | 1 (1)
Vesicoureteric reflux (Renal and urinary disorders) | 1 (1) | 0 (0)
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 (1) | 0 (0)
Bladder neck sclerosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 3 (3) | 2 (2)
Diabetic nephropathy (Renal and urinary disorders) | 10 (12) | 26 (38)
Renal impairment (Renal and urinary disorders) | 2 (2) | 4 (4)
Chronic kidney disease (Renal and urinary disorders) | 2 (2) | 6 (6)
Urethral stenosis (Renal and urinary disorders) | 1 (1) | 2 (2)
Stress urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 38 (39) | 46 (48)
Lower urinary tract symptoms (Renal and urinary disorders) | 0 (0) | 1 (1)
End stage renal disease (Renal and urinary disorders) | 0 (0) | 2 (3)
Ureterolithiasis (Renal and urinary disorders) | 6 (7) | 5 (6)
Subacute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 12 (12) | 10 (10)
Breast mass (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Breast necrosis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Endometrial hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 2 (2)
Prostatic disorder (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Prostatism (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 1 (1) | 3 (3)
Uterine polyp (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Prostatomegaly (Reproductive system and breast disorders) | 1 (1) | 2 (2)
Female genital tract fistula (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Scrotal dermatitis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (5)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 12 (12) | 9 (10)
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 5 (5)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 22 (24) | 16 (26)
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 (11) | 9 (10)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (5)
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 7 (10)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (6)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 11 (11)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (6)
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 9 (12)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 4 (5)
Pharyngeal mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Laryngeal disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hepatic hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Alveolar lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lung perforation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Small airways disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Angioedema (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hidradenitis (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Palmoplantar keratoderma (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pemphigoid (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (4)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Skin necrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 12 (12) | 15 (20)
Neuropathic ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Diabetic ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Necrobiosis lipoidica diabeticorum (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Diabetic foot (Skin and subcutaneous tissue disorders) | 23 (24) | 18 (22)
Angiokeratoma (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Reactive perforating collagenosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Diabetic cheiroarthropathy (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Abscess drainage (Surgical and medical procedures) | 0 (0) | 3 (3)
Aortic aneurysm repair (Surgical and medical procedures) | 1 (1) | 1 (1)
Aortic valve replacement (Surgical and medical procedures) | 1 (1) | 1 (1)
Appendicectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Arteriovenous fistula operation (Surgical and medical procedures) | 2 (2) | 0 (0)
Bladder calculus removal (Surgical and medical procedures) | 1 (1) | 0 (0)
Bladder neck resection (Surgical and medical procedures) | 0 (0) | 1 (1)
Cardiac pacemaker insertion (Surgical and medical procedures) | 1 (1) | 0 (0)
Carotid endarterectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Cholecystectomy (Surgical and medical procedures) | 2 (2) | 7 (7)
Circumcision (Surgical and medical procedures) | 1 (1) | 0 (0)
Coronary artery bypass (Surgical and medical procedures) | 1 (1) | 1 (1)
Finger amputation (Surgical and medical procedures) | 1 (1) | 0 (0)
Foot amputation (Surgical and medical procedures) | 1 (1) | 0 (0)
Hip arthroplasty (Surgical and medical procedures) | 4 (4) | 2 (2)
Hysterectomy (Surgical and medical procedures) | 2 (2) | 1 (1)
Incisional hernia repair (Surgical and medical procedures) | 0 (0) | 1 (1)
Inguinal hernia repair (Surgical and medical procedures) | 0 (0) | 2 (2)
Insertion of ambulatory peritoneal catheter (Surgical and medical procedures) | 0 (0) | 1 (1)
Intensive care (Surgical and medical procedures) | 0 (0) | 1 (1)
Internal fixation of fracture (Surgical and medical procedures) | 1 (1) | 0 (0)
Knee arthroplasty (Surgical and medical procedures) | 8 (8) | 9 (9)
Leg amputation (Surgical and medical procedures) | 3 (3) | 5 (5)
Lipoma excision (Surgical and medical procedures) | 0 (0) | 1 (1)
Lung lobectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Nasal polypectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Parathyroidectomy (Surgical and medical procedures) | 1 (1) | 1 (1)
Parotidectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Radical hysterectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Radioactive iodine therapy (Surgical and medical procedures) | 0 (0) | 1 (1)
Removal of foreign body from larynx (Surgical and medical procedures) | 0 (0) | 1 (1)
Removal of internal fixation (Surgical and medical procedures) | 2 (2) | 0 (0)
Renal cyst excision (Surgical and medical procedures) | 0 (0) | 1 (1)
Renal stone removal (Surgical and medical procedures) | 2 (3) | 0 (0)
Roux loop conversion (Surgical and medical procedures) | 3 (3) | 0 (0)
Scar excision (Surgical and medical procedures) | 1 (1) | 0 (0)
Skin ulcer excision (Surgical and medical procedures) | 0 (0) | 1 (2)
Spinal decompression (Surgical and medical procedures) | 1 (1) | 0 (0)
Spinal laminectomy (Surgical and medical procedures) | 3 (3) | 1 (1)
Toe amputation (Surgical and medical procedures) | 4 (4) | 3 (3)
Transurethral prostatectomy (Surgical and medical procedures) | 2 (2) | 4 (4)
Umbilical hernia repair (Surgical and medical procedures) | 0 (0) | 1 (1)
Uterine polypectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Vitrectomy (Surgical and medical procedures) | 3 (3) | 2 (3)
Implantable defibrillator insertion (Surgical and medical procedures) | 0 (0) | 1 (1)
Knee operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Shoulder arthroplasty (Surgical and medical procedures) | 1 (1) | 0 (0)
Coronary revascularisation (Surgical and medical procedures) | 0 (0) | 1 (1)
Ureteral stent insertion (Surgical and medical procedures) | 0 (0) | 1 (1)
Radical prostatectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Diabetes mellitus management (Surgical and medical procedures) | 2 (3) | 0 (0)
Preoperative care (Surgical and medical procedures) | 0 (0) | 1 (1)
Transurethral bladder resection (Surgical and medical procedures) | 1 (2) | 1 (1)
Neurolysis (Surgical and medical procedures) | 1 (1) | 0 (0)
Polypectomy (Surgical and medical procedures) | 2 (2) | 3 (3)
Caecum operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Intervertebral disc operation (Surgical and medical procedures) | 2 (2) | 4 (4)
Peripheral artery angioplasty (Surgical and medical procedures) | 2 (2) | 1 (1)
Peripheral nerve decompression (Surgical and medical procedures) | 1 (1) | 0 (0)
Skin neoplasm excision (Surgical and medical procedures) | 1 (1) | 1 (1)
Proctocolectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Cardiac ablation (Surgical and medical procedures) | 1 (1) | 0 (0)
Brachytherapy (Surgical and medical procedures) | 1 (1) | 0 (0)
Limb operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Aortic surgery (Surgical and medical procedures) | 0 (0) | 1 (1)
Bone operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Chemotherapy (Surgical and medical procedures) | 2 (5) | 0 (0)
Colectomy (Surgical and medical procedures) | 3 (3) | 0 (0)
Eye operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Eyelid operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Prostatectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Gastrectomy (Surgical and medical procedures) | 1 (1) | 1 (1)
Gastric bypass (Surgical and medical procedures) | 3 (3) | 2 (2)
Hydrocele operation (Surgical and medical procedures) | 0 (0) | 1 (2)
Lithotripsy (Surgical and medical procedures) | 1 (1) | 0 (0)
Retinal operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Thyroidectomy (Surgical and medical procedures) | 1 (1) | 1 (1)
Tooth extraction (Surgical and medical procedures) | 0 (0) | 1 (1)
Varicose vein operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Skin graft (Surgical and medical procedures) | 1 (1) | 0 (0)
Spinal operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Drug therapy (Surgical and medical procedures) | 1 (1) | 0 (0)
Vascular stent insertion (Surgical and medical procedures) | 1 (1) | 0 (0)
Cataract operation (Surgical and medical procedures) | 7 (9) | 3 (5)
Rectocele repair (Surgical and medical procedures) | 0 (0) | 1 (1)
Percutaneous coronary intervention (Surgical and medical procedures) | 1 (1) | 0 (0)
Intraocular lens implant (Surgical and medical procedures) | 1 (1) | 0 (0)
Neurosurgery (Surgical and medical procedures) | 0 (0) | 1 (1)
Pancreatic stent placement (Surgical and medical procedures) | 1 (1) | 0 (0)
Peripheral artery bypass (Surgical and medical procedures) | 2 (2) | 0 (0)
Large intestinal polypectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Breast conserving surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
Transcatheter aortic valve implantation (Surgical and medical procedures) | 0 (0) | 1 (1)
Metabolic surgery (Surgical and medical procedures) | 2 (2) | 0 (0)
Atrial appendage closure (Surgical and medical procedures) | 1 (1) | 0 (0)
Cheilectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Biliary catheter removal (Surgical and medical procedures) | 1 (1) | 0 (0)
Renal disorder prophylaxis (Surgical and medical procedures) | 0 (0) | 1 (1)
Ocular stem cell transplant (Surgical and medical procedures) | 1 (1) | 0 (0)
Drug delivery device placement (Surgical and medical procedures) | 0 (0) | 1 (1)
Aortic aneurysm (Vascular disorders) | 4 (4) | 1 (1)
Aortic dissection (Vascular disorders) | 1 (1) | 0 (0)
Aortic stenosis (Vascular disorders) | 5 (5) | 2 (2)
Aortitis (Vascular disorders) | 1 (1) | 0 (0)
Arterial thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Circulatory collapse (Vascular disorders) | 1 (1) | 1 (1)
Essential hypertension (Vascular disorders) | 0 (0) | 2 (2)
Giant cell arteritis (Vascular disorders) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 12 (12) | 22 (28)
Hypertensive crisis (Vascular disorders) | 2 (2) | 6 (6)
Hypotension (Vascular disorders) | 2 (2) | 3 (3)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 5 (5)
Peripheral vascular disorder (Vascular disorders) | 0 (0) | 2 (2)
Phlebitis (Vascular disorders) | 1 (1) | 0 (0)
Shock (Vascular disorders) | 0 (0) | 1 (1)
Subclavian steal syndrome (Vascular disorders) | 0 (0) | 1 (1)
Systolic hypertension (Vascular disorders) | 0 (0) | 1 (1)
Thrombophlebitis (Vascular disorders) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 2 (2)
Varicose ulceration (Vascular disorders) | 1 (1) | 0 (0)
Varicose vein (Vascular disorders) | 1 (2) | 0 (0)
Vasculitis (Vascular disorders) | 1 (1) | 0 (0)
Post thrombotic syndrome (Vascular disorders) | 1 (1) | 0 (0)
Labile hypertension (Vascular disorders) | 0 (0) | 1 (1)
Dry gangrene (Vascular disorders) | 1 (1) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 3 (3) | 5 (5)
Peripheral artery aneurysm (Vascular disorders) | 0 (0) | 1 (1)
Peripheral artery occlusion (Vascular disorders) | 2 (2) | 2 (2)
Hypertensive emergency (Vascular disorders) | 2 (3) | 3 (3)
Hypertensive urgency (Vascular disorders) | 1 (1) | 4 (5)
Extremity necrosis (Vascular disorders) | 4 (4) | 1 (1)
Peripheral embolism (Vascular disorders) | 1 (1) | 0 (0)
Diabetic vascular disorder (Vascular disorders) | 1 (1) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 2 (2) | 6 (7)
Subclavian artery occlusion (Vascular disorders) | 1 (1) | 0 (0)
Peripheral artery stenosis (Vascular disorders) | 1 (1) | 1 (1)
Peripheral artery thrombosis (Vascular disorders) | 1 (1) | 1 (1)
Peripheral artery aneurysm rupture (Vascular disorders) | 0 (0) | 1 (1)
Device malfunction (Product Issues) | 0 (0) | 1 (1)
Device loosening (Product Issues) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Finerenone (N=3683) | Placebo (N=3658)
Anaemia (Blood and lymphatic system disorders) | 210 (227) | 199 (215)
Constipation (Gastrointestinal disorders) | 185 (213) | 171 (192)
Diarrhoea (Gastrointestinal disorders) | 235 (283) | 220 (271)
Oedema peripheral (General disorders) | 197 (227) | 278 (343)
Bronchitis (Infections and infestations) | 191 (238) | 176 (214)
Nasopharyngitis (Infections and infestations) | 318 (537) | 327 (497)
Upper respiratory tract infection (Infections and infestations) | 225 (351) | 203 (310)
Urinary tract infection (Infections and infestations) | 246 (335) | 220 (313)
Hyperkalaemia (Metabolism and nutrition disorders) | 322 (470) | 159 (219)
Arthralgia (Musculoskeletal and connective tissue disorders) | 296 (379) | 260 (337)
Back pain (Musculoskeletal and connective tissue disorders) | 260 (288) | 252 (287)
Dizziness (Nervous system disorders) | 190 (218) | 166 (184)
Hypertension (Vascular disorders) | 199 (241) | 296 (347)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2019-03-12): https://cdn.clinicaltrials.gov/large-docs/49/NCT02545049/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-15): https://cdn.clinicaltrials.gov/large-docs/49/NCT02545049/SAP_001.pdf